CLINICAL TRIAL: NCT01446562
Title: Phase II Trial of Y90 Ibritumomab Tiuxetan Post Rituximab-Cyclophosphamide, Doxobrubicn, Vincristine and Prednisone (R-CHOP) Chemotherapy for Newly Diagnosed Patients With Advanced Stage Follicular Lymphoma
Brief Title: Y90 Ibritumomab Tiuxetan Post R-CHOP Chemotherapy for Advanced Stage Follicular Lymphoma
Acronym: ZEVISS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Neil Berinstein, Medical Oncologist, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZEVISS
Record Dates: First submitted 2011-08-11; First posted 2011-10-05 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Y90 Ibritumomab Tiuxetan (Experimental): Addition of Y90 Ibritumomab Tiuxetan RIT to CHOP-R treatment for follicular lymphoma-patients also receive maintenance Rituximab every 3 months for 2 years after the Y90 Ibritumomab Tiuxetan
  Interventions: Biological: Y90 Ibritumomab Tiuxetan RIT

INTERVENTIONS:
Biological: Y90 Ibritumomab Tiuxetan RIT — 40 mCi/kg
  Other Names: Zevalin

SUMMARY:
The primary objective of this study is to establish in a prospective phase II study the efficacy of 90Yttrium ibritumomab tiuxetan (90Y-RIT) after first line induction immuno-chemotherapy with R-CHOP in patients with high-risk advanced stage follicular non-Hodgkin's lymphoma, as assessed by the complete response rate.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, open label, single-centre phase II trial of R-CHOP followed by 90Y-RIT in patients with previously untreated, high-risk, advanced stage follicular non-Hodgkin's lymphoma.

Patients who meet all inclusion criteria (and no exclusion criteria) will receive first line treatment with the R-CHOP regimen. R-CHOP comprises rituximab 375 milligrams per square meter (mg/m2) intravenously (IV), cyclophosphamide 750mg/m2 IV, doxorubicin 50mg/m2 IV, and vincristine 1.4mg/m2 IV (to a maximum dose of 2.0mg) on day 1 and prednisone 100mg per os (po) daily for 5 days. Treatment cycles will be repeated every 3 weeks for a total of 6 cycles. Patients will be evaluated for response according to the after 3 and 6 cycles of R-CHOP (see response definitions below).

Dose modifications for non-hematologic and hematologic adverse events will be guided by NCI Common Terminology Criteria for Adverse Events Version 3.0 (CTCAE). After 3 cycles of R-CHOP, patients with disease progression will go off study while responders will continue with further treatment. Patients with stable disease can continue on the protocol or discontinue the study, as decided by the treating physician. Final response evaluation to R-CHOP induction will take place 4-6 weeks after the 6th cycle. Patients with disease progression will go off study, while those with stable disease and evidence of response will be eligible for post-induction 90Y-RIT.

Post-induction 90Y-RIT will be administered within 4-8 weeks of completion of the R-CHOP regimen. Patients must meet criteria for administration of 90Y-RIT therapy, including: (1) achievement of at least stable disease determined 4-6 weeks after the completion of R-CHOP therapy; (2) repeat bone marrow investigation confirming less than 25% marrow involvement with follicular lymphoma; and (3) platelet count greater than or equal to 100,000/mm3. Eligible patients will receive an infusion of rituximab 250mg/m2 on day 1 followed a week later (day 8) by an additional dose of rituximab and a single dose of 90Y ibritumomab tiuxetan at a dose of 0.4 milliCurries per kilogram (mCi/kg) for patients with a platelet count ≥150,000/mm3 or 0.3 mCi/kg for patients with platelets <150,000/cubic millimeter (mm3). The maximum dose regardless of weight will be 32 mCi. Dosimetry and imaging studies for biodistribution will not be mandated in this protocol.

The primary endpoint for the study is the final complete response (CR) rate, defined according to International Working Group criteria, and measured 3 months after completion of the treatment (measured from day 1 of the 90Y-RIT therapy). Hence, CR implies the elimination of all lymphoma manifestations including complete disappearance of all detectable clinical and radiographic evidence of disease and all disease-related symptoms if present before therapy.

Secondary outcomes include the determination of overall and partial response (PR) rates and the conversion of partial responses/stable disease to complete responses. A subset of patients (with pre-treatment polymerase chain reaction (PCR) analysis positive for the characteristic t(14;18)(q32;q21) B Cell Lymphoma-2 gene/Immunoglobulin Heavy chain (BCL2/IGH) translocation associated with follicular lymphoma) will be monitored by quantitative PCR for minimal residual disease and will have molecular remission rates documented (conversion from PCR positive to negative). Time-to-event outcomes will include time-to-treatment failure, time to progression, and overall survival. The frequency and severity of side effects will be recorded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events Version 3.0 (CTCAE). The safety and tolerability of the study drugs will be evaluated by relevant laboratory parameters at 2 week intervals during the induction chemotherapy and following the administration of 90Y ibritumomab tiuxetan until the final response assessment (3 months after the radioimmunoconjugate dose). Thereafter, these parameters will be repeated quarterly for the first 2 years, and at any restaging visit thereafter. Long-term adverse events include the development of myelodysplastic syndrome and acute myeloid leukemia, other secondary cancers.

Immunoquantitation and vaccine-specific immunity (serology) will also be assayed during the long-term follow-up period.

The study is expected to accrue over a 24-month period. The time-to-event outcomes will continue to be assessed in the follow-up period, scheduled to end 2 years after the last patient has received 90Y-RIT. Restaging will be carried out after 3 and 6 cycles of the R-CHOP induction therapy, and 3 months after the administration of 90Y-RIT (final response assessment). Thereafter, restaging will be carried out every 6 months until completion of the 2 year follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years.
* Biopsy demonstration of a CD20+ follicular non-Hodgkin's lymphoma diagnosed according to the World Health Organization (WHO) classification (grade I, II, or IIIa).
* Staging demonstration of advanced stage disease (stage III or IV) according to the Ann Arbor staging system.
* Intermediate or high-risk prognostic score (2-5 points) according to the follicular lymphoma international prognostic index (FLIPI).
* Adequate performance status (less than or equal to 2) according to the Eastern Cooperative Oncology Group (ECOG) (Zubrod) scale.
* No prior radiotherapy or systemic therapy, including chemotherapy or immunotherapy (rituximab).
* Bi-dimensional measurable disease by physical examination or radiographic evaluation (disease measurements at least 1.5 cm x 1.5 cm) or assessable disease on bone marrow evaluation.
* Clinical criteria for therapeutic intervention, as previously reported by Hiddeman, including one of: the presence of B-symptoms, bulky disease (mediastinal lymphomas >7.5 cm or other lymphomas >5 cm in maximal diameter), an impairment of normal hematopoesis with hemoglobin <10g/mm3, granulocytes <1500/mm3, or platelets <100,000/mm3, and/or a rapidly progressive disorder.
* Patient consent must be obtained according to the Sunnybrook Health Sciences Centre Research Ethics Board requirements. A sample consent form is given in Appendix I. The patient must sign the consent form prior to registration.
* Patients must be accessible for treatment and follow up. Patients registered on this trial must complete their therapy with 90Y Ibritumomab Tiuxetan at the participating centre. Induction chemotherapy with R-CHOP should also be completed at the participating centre, but exceptions can be made according to the discretion of the centre's primary investigator.
* Protocol treatment is to begin within 5 working days of patient registration

Exclusion Criteria:

* Pregnancy or women who intend to breast-feed during the study period.
* Follicular non-Hodgkin's lymphoma grade IIIb histology, according to the World Health Organization (WHO) classification.
* Known human immunodeficiency virus infection or hepatitis B viral infection.
* Life expectancy less than or equal to 3 months, according to physician judgement.
* Evidence of left ventricular (LV) dysfunction (ejection fraction less than or equal to 50%). Demonstration of LV function is required in patients over the age of 60 or in patients with a prior history of hypertension, congestive heart failure, peripheral vascular disease, cerebrovascular disease, coronary artery disease, or cardiac arrhythmia.
* Serum creatinine, alkaline phosphatase, or total bilirubin >2.5 times the upper limit of the normal value, unless clearly related to lymphoma.
* Concurrent uncontrolled medical disease, including severe congestive heart failure, myocardial infarction within 6 months prior to enrollment, severe chronic renal failure, or active infection, with the severity of disease judged according to the discretion of the treating physician.
* Patients with a history of other malignancies, except: (1) adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or (2) other solid tumours curatively treated with no evidence of disease for > 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2007-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
The primary endpoint for this study is the complete response rate measured 3 months after the dose of 90Y-RIT | 3 months after the dose of 90Y-RIT
  The primary endpoint for the study is the final complete response (CR) rate, defined according to International Working Group criteria 24, and measured 3 months after completion of the treatment (measured from day 1 of the 90Y-RIT therapy). Hence, CR implies the elimination of all lymphoma manifestations including complete disappearance of all detectable clinical and radiographic evidence of disease and all disease-related symptoms if present before therapy.

SECONDARY OUTCOMES:
toxicities | entry into trial until 6 weeks post 90Y ibritumomab tiuxetan treatment (week 30)
  Toxicity associated with R-CHOP induction and 90Y ibritumomab tiuxetan treatment will be assessed by monitoring the incidence, severity, and type of adverse events. Adverse events will be recorded according to the NCI CTCAE . In addition, changes in physical examination findings, vital signs, and clinical laboratory results (complete blood count, differential, and chemistry) will be documented.
Conversion of partial responses to complete responses | 6 weeks post 90Y ibritumomab tiuxetan treatment
  CTT assessment before and after 90Y ibritumomab tiuxetan treatment - Bone marrow aspiration and biopsies in those patients with positive Bone marrows prior to 90Y ibritumomab tiuxetan treatment.
Minimal residual disease | For two years post study entry
  Peripheral blood will be assessed every 6 months for the two years from entry into the trial and subjected to PCR analysis for evidence of lymphoma cells with the t(14;18)
Time to treatment failure | Two years of the study duration
  Evidence of progression will be assessed every 6 months for two years from study entry clinically and radiologically to determine the date of disease progression
Overall survival | two years of study duration
  Survival will be assessed continually throughout the two year study period

CONTACTS AND LOCATIONS:
Overall Officials: Neil L Berinstein, MD, FRCP(C), Principal Investigator — Sunnybrook Health Sciences Centre, Odette Cancer Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Odette Cancer Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Berinstein NL, Pennell NM, Weerasinghe R, Buckstein R, Piliotis E, Imrie KR, Chodirker L, Cussen MA, Miles E, Reis MD, Ghorab Z, Cheung MC. Management of newly diagnosed high-risk and intermediate-risk follicular lymphoma with 90 Y ibritumomab tiuxetan in a phase II study. Hematol Oncol. 2018 Apr 30. doi: 10.1002/hon.2513. Online ahead of print. PMID 29709062